CLINICAL TRIAL: NCT03082378
Title: Central Obesity and the Prognosis of Hepatocellular Carcinoma After Microwave Ablation
Brief Title: Central Obesity and Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu Jie, Professor, Chinese PLA General Hospital
Other Study IDs: 301jrcsk
Record Dates: First submitted 2017-03-12; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Hepatocellular Carcinoma; Obesity; Microwave Ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recurrence and metastases after microwave ablation(MWA) of hepatocellular carcinoma(HCC) are the major factors that influence the survival. Obesity has been reported was significantly correlated with increased risk of developing HCC.

In this study, we will analysis the association of multiple obesity index(waist circumference,waist-hip ratio and body mass index) with the prognosis of HCC treated by MWA.

ELIGIBILITY:
Inclusion Criteria:

* absence of ascites or the depth of ascites on US detection less than 4 cm;
* a normal serum total bilirubin level or less than 60 µmol/L;
* a normal albumin level or not less than 30 g/L;
* for radical treatment, single lesion of 8 cm or smaller, three or fewer multiple lesions with a maximum diameter of 4 cm or less, absence of portal vein cancerous thrombus or extrahepatic metastases;
* for palliative treatment, those with large or multiple lesions, suffering multiple metastases and unsuitable for other modalities can be considered to undergo the MWA on the condition of good hepatic function and blood coagulation function to tolerate the procedure.

Exclusion Criteria:

1. clinical evident liver failure, such as massive ascites or hepatic encephalopathy or with a trance-like state
2. severe blood coagulation dysfunction (prothrombin time of more than 30 seconds, prothrombin activity less than 40%, and platelet count less than 30 cells×109/L)
3. high intrahepatic tumor burden (tumor volume >70% of the target liver volume or multiple tumor nodules) or high extrahepatic tumor burden
4. acute or active inflammatory and infectious lesions at any organ
5. acute or severe chronic renal failure, pulmonary insufficiency or heart dysfunction
6. relative contraindication concerns medical risk for the tumor proximity to diaphragm, gastrointestinal tract, gallbladder, pancreas, hepatic hilum and major bile duct or vessels, which may require adjunctive techniques to prevent off-target heating of adjacent structures during the ablation procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HCC patients are treated by ultrasound-guided percutaneous MWA
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
survival | 3 years
  Percentage of participants who survived up to end time point as assessed by Kaplan-Meier

SECONDARY OUTCOMES:
intra-hepatic metastasis | 3 years
  Percentage of participants who present metastasis in the liver up to end time point as assessed by Kaplan-Meier
extra-hepatic metastasis | 3 years
  Percentage of participants who present metastasis outside the liver up to end time point as assessed by Kaplan-Meier
local tumor progression | 3 years
  Percentage of participants who present tumor progression around the ablation zone up to end time point as assessed by Kaplan-Meier
complication | 3 years
  number of participants with side effect and major complication

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yu, Dr, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No